CLINICAL TRIAL: NCT01029886
Title: Safety and Efficacy of Exenatide Once Weekly Versus Liraglutide in Subjects With Type 2 Diabetes and Inadequate Glycemic Control Treated With Lifestyle Modification and Oral Antidiabetic Medications
Brief Title: Safety and Efficacy of Exenatide Once Weekly Versus Liraglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWDE
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; liraglutide; Victoza; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide once weekly
- 2 (Active Comparator)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2mg, once weekly
  Arms: 1
Drug: liraglutide — subcutaneous injection, forced titration to 1.8mg, once daily
  Other Names: Victoza
  Arms: 2

SUMMARY:
No head to head comparisons between exenatide once weekly and liraglutide have been performed. Therefore, the purpose of this study is to compare exenatide once weekly to once-daily liraglutide with regard to HbA1c, body weight, subject-reported outcomes, and other clinical benefits. The study includes a 26-week treatment period and a safety follow-up visit 10 weeks after the final study drug dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Have suboptimal glycemic control as evidenced by an HbA1c measurement at study start 7.1% and 11.0%, inclusive
* Have a body mass index (BMI) ≤45 kg/m^2
* Have been treated with lifestyle modification (diet and exercise) and with one of the following single oral antidiabetic agents (OADs) or combinations of OADs administered at maximum tolerated dose:

  * metformin
  * SU
  * metformin plus an SU
  * metformin plus pioglitazone

Exclusion Criteria:

* Have any contraindication, allergy, or hypersensitivity for the study drug (exenatide once weekly or liraglutide), exenatide twice daily, the OAD(s) being used, or the excipients contained in these agents
* If taking metformin and have a contraindication to metformin use
* Have been treated within 8 weeks of study start with systemic glucocorticoid therapy by oral, intravenous, intra-articular, or intramuscular route
* Have been treated with drugs that promote weight loss (e.g., Xenical® [orlistat], Meridia® [sibutramine], Acomplia® [rimonabant], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of study start
* Have taken any of the following excluded medications for more than 1 week within the 3 months prior to study start, or have taken any of the following excluded medications within 1 month prior to study start:

  * Insulin
  * Alpha-glucosidase inhibitors (e.g., Glyser® [miglitol] or Precose® [acarbose])
  * Meglitinides (e.g., Prandin® [repaglinide] or Starlix® [nateglinide])
  * Avandia® (rosiglitazone)
  * Dipeptidyl peptidase (DPP)-4 inhibitors (e.g., Januvia™ [sitagliptin], Galvus® [vildagliptin], Onglyza™ [saxagliptin])
  * Symlin® (pramlintide acetate)
* Have donated blood within 30 days prior to study start or have had a blood transfusion or severe blood loss within 3 months prior to study start
* Have at any time, including a clinical trial, taken exenatide once weekly, exenatide twice daily, liraglutide, or any other GLP-1 receptor agonist or GLP-1 analog
* Are currently enrolled in, or discontinued within the last 3 months or longer if required by local guidelines, from a clinical trial involving use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously been screen-failed from this study for any reason
* If a subject discontinues metformin, sulfonylurea, or pioglitazone prior to screening, the subject can be included if they discontinued the medication (whether alone or as component of combined medication) according to a specific schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (108):
- Argentina (3):
  - Research Site, Buenos Aires
  - Research site, Mendoza
  - Research Site, Rosario
- Australia (3):
  - Research Site, Box Hill
  - Research Site, Geelong
  - Research Site, Keswick
- Research Site, Vienna, Austria
- Belgium (5):
  - Research site, Bonheiden
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Leuven
  - Research Site, Liège
- Canada (8):
  - Research Site, Charlottetown
  - Research Site, Gatineau
  - Research Site, Ottawa
  - Research Site, Sherbrooke
  - Research Site, Vancouver
  - Research Site, Victoria
  - Research Site, Windsor
  - Research Site, Winnipeg
- Czechia (3):
  - Research Site, Brandýs nad Labem
  - Research Site, Prague
  - Research Site, Přerov
- France (7):
  - Research Site, Grenoble
  - Research Site, Le Creuzot
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Strasbourg
- Germany (13):
  - Research Site, Bad Staffelstein
  - Research Site, Beckum
  - Research Site, Biberach
  - Research Site, Datteln
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Ludwigshafen
  - Research Site, Mainz
  - Research Site, Meissen
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Riesa
  - Research Site, Stuttgart
- Greece (3):
  - Research Site, Athens
  - Research Site, Cholargós
  - Research Site, Pátrai
- Hungary (6):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Makó
  - Research Site, Mosonmagyaróvár
  - Research Site, Nagykanizsa
  - Research Site, Székesfehérvár
- India (10):
  - Research Site, Aligarh
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Coimbatore
  - Research Site, Hyderabad
  - Research Site, Indore
  - Research Site, Karnal/Haryana
  - Research site, Karnataka
  - Research Site, Mumbai
  - Research Site, Pune
- Israel (4):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Raanana
- Italy (7):
  - Research Site, Bari
  - Research Site, Cagliari
  - Research Site, Catanzaro
  - Research Site, Chieti
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Treviglio
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research site, Rzeszów
  - Research Site, Warsaw
- Romania (4):
  - Research site, Bucharest
  - Research site, Galati
  - Research site, Iași
  - Research site, Oradea
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Malacky
  - Research Site, Martin
- South Africa (5):
  - Research Site, Halfway House
  - Research Site, Johannesburg
  - Research Site, Kempton Park
  - Research Site, Parktown
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (6):
  - Research Site, Alicante
  - Research Site, Alzira
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Teruel
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Xindian
  - Research Site, Yung-Kang, Tainan
  - Research Site, Zhonghe

REFERENCES:
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Buse JB, Nauck M, Forst T, Sheu WH, Shenouda SK, Heilmann CR, Hoogwerf BJ, Gao A, Boardman MK, Fineman M, Porter L, Schernthaner G. Exenatide once weekly versus liraglutide once daily in patients with type 2 diabetes (DURATION-6): a randomised, open-label study. Lancet. 2013 Jan 12;381(9861):117-24. doi: 10.1016/S0140-6736(12)61267-7. Epub 2012 Nov 7. PMID 23141817

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide Once Daily: Subcutaneous injection, forced titration to 1.8mg, once daily
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Started | 461 | 451
Intent to Treat (ITT) | 461 | 450
Completed | 400 | 391
Not Completed | 61 | 60
Not completed — Adverse Event | 12 | 25
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 6
Not completed — Protocol Violation | 17 | 5
Not completed — Withdrawal by Subject | 8 | 18
Not completed — Entry Criteria Not Met | 13 | 5
Not completed — Sponsor Decision | 1 | 0
Not completed — Loss Glucose Control | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily | Total
Number analyzed (Participants) | 461 | 450 | 911
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 386 | 360 | 746
  >=65 years | 75 | 90 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.43) | 56.7 (9.59) | 56.6 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 205 | 412
  Male | 254 | 245 | 499
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.45 (1.014) | 8.43 (0.996) | 8.44 (1.004)
Weight [Mean (Standard Deviation); unit: kg] | 90.88 (19.472) | 91.13 (19.118) | 91.00 (19.288)
Background Oral Antidiabetic Agent (OAD) [Number; unit: participants]
  Metformin (MET) | 150 | 136 | 286
  Sulfonylurea (SU) | 18 | 18 | 36
  Pioglitazone (PIO) | 1 | 0 | 1
  MET+SU | 275 | 277 | 552
  MET+PIO | 16 | 18 | 34
  MET+SU+PIO | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population: all patients who were randomized and received study drug. All observed data from all scheduled visits (including early termination visits) were included in the mixed-model repeated measures (MMRM) analysis. Data collected at the early termination visits were mapped into the following scheduled visits.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 390 | 386
percentage of total hemoglobin | -1.28 (0.05) | -1.48 (0.05)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; A sample of 408 subjects in each treatment arm would provide approximately 90% power to detect a true difference between treatments of 0.25% in change in HbA1c from baseline with a 2 sided t-test at a significance level of 0.05, assuming a common standard deviation of 1.1%. MMRM model includes treatment, baseline HbA1c, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Non-Inferiority or Equivalence — Superiority of exenatide once weekly with respect to change in HbA1c was concluded if the upper limit of the 2-sided 95% confidence interval (CI) for the treatment difference (exenatide once weekly minus liraglutide) was less than zero. Non-inferiority was concluded if the upper limit of the CI was <0.25%; p = 0.002, Mixed Models Analysis; Least Squares Mean Difference = 0.21, 95% CI 2-sided [0.08 to 0.33], Standard Error of Mean 0.07

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <7.0% at Week 26
Description: Percentage of patients achieving HbA1c <7.0% at treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population. Missing data at endpoint was imputed using last observation carried forward approach.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 461 | 450
percentage of patients | 52.7 | 60.2
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; Percentage of patients achieving HbA1c <7.0% at Week 26 were compared between treatments using a Cochran-Mantel-Haenszel test, in which HbA1c stratum, country, and background OAD served as stratification factors; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change in Fasting Serum Glucose From Baseline to Week 26
Description: Change in fasting serum glucose from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: ITT Population. All observed data from all scheduled visits (including early termination visits) were included in the MMRM analysis. Data collected at the early termination visits were mapped into the following scheduled visits.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 403 | 385
mmol/L | -1.76 (0.11) | -2.12 (0.12)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline fasting serum glucose, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis; Least Squares Mean Difference = 0.36, 95% CI 2-sided [0.05 to 0.66], Standard Error of Mean 0.15

4. Secondary Outcome: Change in Body Weight From Baseline to Week 26
Description: Change in body weight from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 404 | 398
kg | -2.68 (0.18) | -3.57 (0.18)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline body weight, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Least Squares Mean Difference = 0.90, 95% CI 2-sided [0.39 to 1.40], Standard Error of Mean 0.26

5. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 26
Description: Change in total cholesterol from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 402 | 386
mmol/L | -0.06 (0.04) | -0.15 (0.04)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline total cholesterol, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis; Least Squares Mean Difference = 0.09, 95% CI 2-sided [-0.01 to 0.19], Standard Error of Mean 0.05

6. Secondary Outcome: Change in High-Density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: Change in HDL-C from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 402 | 386
mmol/L | 0.02 (0.01) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline HDL-C, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p = 0.832, Mixed Models Analysis; Least Squares Mean Difference = 0.00, 95% CI 2-sided [-0.02 to 0.02], Standard Error of Mean 0.01

7. Secondary Outcome: Ratio of Fasting Triglycerides at Week 26 to Baseline
Description: Ratio of fasting triglycerides (measured in mmol/L) treatment endpoint at Week 26 to baseline. Log(Postbaseline fasting triglycerides) - log(Baseline fasting triglycerides); change from baseline to the treatment endpoint at Week 26 is presented as ratio of Week 26 to baseline.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 395 | 385
ratio | 0.97 (0.02) | 0.89 (0.02)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; Fasting triglycerides were logarithm-transformed and the change at Week 26 to baseline, expressed as the ratio, was analyzed using a MMRM model with treatment, baseline fasting triglycerides, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Least Squares Mean Difference = 1.09, 95% CI 2-sided [1.04 to 1.15], Standard Error of Mean 0.03

8. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26
Description: Change in SBP from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 404 | 398
mmHg | -2.48 (0.56) | -3.45 (0.57)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline SBP, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p = 0.205, Mixed Models Analysis; Least Squares Mean Difference = 0.97, 95% CI 2-sided [-0.53 to 2.47], Standard Error of Mean 0.76

9. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Week 26
Description: Change in DBP from baseline to the treatment endpoint at Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Number analyzed (Participants) | 404 | 398
mmHg | -0.49 (0.37) | -0.51 (0.37)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Liraglutide Once Daily; MMRM model includes treatment, baseline DBP, HbA1c stratum, country, background OAD, week of visit, and treatment-by-week interaction as fixed effects and subject and error as random effects; Test type: Superiority or Other; p = 0.981, Mixed Models Analysis; Least Squares Mean Difference = 0.01, 95% CI 2-sided [-0.96 to 0.98], Standard Error of Mean 0.50

10. Secondary Outcome: Assessment of Event Rate of Treatment-emergent Hypoglycemic Events
Description: Major hypoglycemia: any episode with symptoms consistent with hypoglycemia that resulted in loss of consciousness or seizure with prompt recovery in response to administration of glucagon or glucose OR documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) and required the assistance of another person. Minor hypoglycemia: any sign or symptom associated with hypoglycemia that is either self-treated by the patient or resolves on its own AND has a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia. Event rate per subject year was calculated for each subject: (number of events observed from a subject/exposure from a subject)*365.25 where exposure = last post-baseline visit date - baseline visit date. Mean and Standard Error were then derived from ITT.
Time Frame: Baseline to Week 26
Population: ITT Population.
Measure: Mean (Standard Error); unit: events per subject-year
Groups:
- Exenatide Once Weekly With SU Use at Screening: Subcutaneous injection, 2mg, once weekly and with SU use at screening
- Liraglutide Once Daily With SU Use at Screening: Subcutaneous injection, forced titration to 1.8mg, once daily and with SU use at screening
- Exenatide Once Weekly Without SU Use at Screening: Subcutaneous injection, 2mg, once weekly and without SU use at screening
- Liraglutide Once Daily Without SU Use at Screening: Subcutaneous injection, forced titration to 1.8mg, once daily and without SU use at screening
Arm/Group | Exenatide Once Weekly With SU Use at Screening | Liraglutide Once Daily With SU Use at Screening | Exenatide Once Weekly Without SU Use at Screening | Liraglutide Once Daily Without SU Use at Screening
Number analyzed (Participants) | 294 | 296 | 167 | 154
events per subject-year
  Major Hypoglycemia | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Minor Hypoglycemia | 0.76 (0.143) | 0.55 (0.126) | 0.67 (0.417) | 0.05 (0.026)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Liraglutide Once Daily
Serious Adverse Events (participants affected / at risk) | 13/461 | 7/450
Other Adverse Events (participants affected / at risk) | 160/461 | 212/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=461) | Liraglutide Once Daily (N=450)
Appendicitis (Infections and infestations) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=461) | Liraglutide Once Daily (N=450)
Injection site nodule (General disorders) | 48 | 5
Nausea (Gastrointestinal disorders) | 43 | 93
Nasopharyngitis (Infections and infestations) | 31 | 32
Diarrhoea (Gastrointestinal disorders) | 28 | 58
Headache (Nervous system disorders) | 27 | 38
Decreased appetite (Metabolism and nutrition disorders) | 17 | 29
Vomiting (Gastrointestinal disorders) | 17 | 47
Dyspepsia (Gastrointestinal disorders) | 11 | 27
Therapeutic response unexpected (General disorders) | 11 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days